CLINICAL TRIAL: NCT01427478
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study, to Evaluate the Efficacy of Afatinib (BIBW2992) in Maintenance Therapy After Post- Operative Radio-chemotherapy in Squamous-cell Carcinoma of the Head and Neck: GORTEC 2010-02
Brief Title: Evaluation of Afatinib in Maintenance Therapy in Squamous Cell Carcinoma of the Head and Neck
Acronym: BIBW2992ORL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIBW2992 ORL; 2010-023265-22 (EudraCT Number)
Record Dates: First submitted 2011-08-31; First posted 2011-09-01 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck squamous cell carcinoma; Post operative radio-chemotherapy; Randomisation; Maintenance treatment; Afatinib
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Afatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AFATINIB (Experimental): Radiotherapy combined with a chemotherapy by Cisplatin IV at the dose of 100mg/m2 every 3 weeks, followed by a maintenance therapy with BIBW 2992 for 1 year at the dose of 40 mg/during the 1st month and then 50 mg/d during the 11 following months
  Interventions: Drug: AFATINIB
- PLACEBO (Placebo Comparator): Radiotherapy associated with a chemotherapy by Cisplatin IV at the dose of 100mg/m2 every 3 weeks, followed by a maintenance therapy with placebo of BIBW 2992 for 1 year at the dose of 40 mg/during the 1st month and then 50 mg/d during the 11 following months
  Interventions: Drug: Placebo of AFATINIB

INTERVENTIONS:
Drug: AFATINIB — AFATINIBat the dose of 40 mg/during the 1st month and then 50 mg/d during the 11 following months
  Other Names: BIBW 2992
  Arms: AFATINIB
Drug: Placebo of AFATINIB — placebo of Afatinib at the dose of 40 mg/during the 1st month and then 50 mg/d during the 11 following months
  Other Names: Placebo of BIBW 2992
  Arms: PLACEBO

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Afatinib in maintenance therapy after post-operative radiochemotherapy (66 Gy and Cisplatin at the dose of 100mg/m2 every 3 weeks)in squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
The reference treatment for operated squamous cell carcinoma of the head and the neck is a radiochemotherapy with Cisplatin (in the dose of intravenous 100 mg / m2 IV) every 3 weeks).

The Receptor of EGFR (Epidermal Growth Factor) or REGF is a membrane receptor; it's activation leads the cellular growth and inhibits apoptotic capacities. This receptor is overexpressed in numerous solid tumors, including ENT tumors. Several clinical studies showed that an over expression of the REGF in ENT tumors was a dominant factor of poor prognostic.

Afatinib (BIBW2992) is a strong and irreversible inhibitor of the EGFR ( type 1 human epidermic growth factor receptor, also known as HER1) and of the HER2 (human epidermal growth factor receptor 2).

Currently, 3 phase III clinical studies in postoperative situation and using an anti-REGF are in progress: 2 in concomitant situation with the radiotherapy and 1 both in concomitance and in adjuvant therapy with radiotherapy.

The preliminary results of a phase II study show that Afatinib is efficient in patients with local or metastatic relapse of a squamous cell carcinoma of the sphere ENT after a first line with Cisplatin and its tolerance is correct.

These data lead us to propose in post-operative situation, in patients with a squamous cell carcinoma of the head and neck, a radiochemotherapy with Cisplatin followed by a treatment of maintenance by Afatinib or by placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically-confirmed diagnosis of non metastatic squamous-cell carcinoma of oral cavity ; oropharynx, larynx or hypopharynx.
* Macroscopically complete resection of disease.
* High-risk histological features defined as :

Microscopically incomplete tumour resection and/or invasion of regional lymph nodes with extracapsular extension (pN+R+)

* Indication of radio-chemotherapy (at least 60 Gy of radiotherapy and at least 2 cycles of chemotherapy)
* Start of radio-chemotherapy within 8 weeks after surgery
* Performance Status (PS) ECOG <= 2
* Adequate Blood tests, renal and liver functions in the 15 days prior inclusion defined as :

Hemoglobin > 9 g/dL Neutrophil count > 1500 x 109/L Platelets > 100 x 109/L Total bilirubin < 1,5x upper limit of normal (ULN) SGOT and SGPT < 2,5 x ULN Alkaline Phosphatase < 2,5 xULN Serum creatinine < 110 µmol/L or creatinine clearance > 55 ml/min (estimated by Cockcroft Formula) Absence of proteinuria

* Women of childbearing age must use adequate means of contraception(oral hormon contraceptive, intrauterine contraceptive device, double barrier method of contraception).
* Mandatory affiliation with a healthy security insurance.
* Dated and signed written informed consent.

Exclusion Criteria:

* Macroscopic residual tumour after resection(R2)
* Metastatic disease
* Prior treatment for Head and neck cancer with chemotherapy, radiotherapy or any cancer target therapy
* Prior or concomitant malignancies (except for basal cell skin cancer ; in situ cervical carcinoma or other malignancies with a complete response > 5 years)
* History of heavy hypersensibility reaction to Cisplatin
* Uncontrolled pulmonary, cardiac , hepatic or renal disease.
* History of interstitial pneumopathy
* Significant cardiovascular disease :

Congestive cardiac failure> New York Heart Association (NYHA) Class II Myocardial infraction within 6 months prior to inclusion Unstable angina Severe cardiac arrythmia Uncontrolled hypertension while receiving appropriate medication (≥ 160 mm Hg systolic and/or ≥ 90 mm Hg diastolic) Disorder of left ventricular function with ejection fraction < 50% Severe cerebrovascular accident within 6 months prior to inclusion History of severe thromboembolism within 6 months prior to inclusion Cardiovascular baseline QTcB >480 ms (Calculated with Bazett Formula) Bradycardia Electrolytic disorders

- Hepatic affection like : hepatitis B or C chronic advanced decompensated hepatitis hepatitic cirrhosis or newly treated chronic hepatitis or nowadays treated with immunosuppressive drugs severe auto-immune hepatitis or disease

* HIV known history
* Recent digestive symptoms with diarrhea as :

Crohn's disease malabsorption syndrome diarrhea Grade CTC ≥ 2

* Active drug or alcohol use or dependence
* Pregnant or breast-feeding women , or no use of effective birth control methods for women of childbearing potential, , or men who don't accept to use an effective birth control methods during the study
* Impossible follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-09; Primary Completion 2020-11 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival 2 years after the end of radiotherapy | 2 years after the end of radiotherapy

SECONDARY OUTCOMES:
Safety profile | Every 28 days during the maintenance therapy,every 2 months during 1 year after maintenance therapy; and every 3 months during the following 3 years
  Safety profile is characterized by type; frequency and seriousness of the toxicities showed by the patients and graded using CTCAE - V04
Quality of life of patient, evaluated by questionnary | Baseline; at the end of radiotherapy, at 1 and 2 years after the beginning of maintenance treatment
  Quality of life will be evaluated at baseline; at the end of radiotherapy and also at 1 and 2 years after the beginning of maintenance treatment. The EORTC's questionnaire QLQ-C30 and the additional module " Head and neck " QLQ-H&N35 will be used.
Overall Survival (OS) | Death
  OS is the time from randomization to the date of death due to any cause or date of the last news.

CONTACTS AND LOCATIONS:
Overall Officials: Séverine RACADOT, MD, Principal Investigator — Centre Léon Bérard, Lyon; Pascal POMMIER, MD, Principal Investigator — Centre Léon Bérard, Lyon
Locations (26):
- France (26):
  - Centre Paul Papin, Angers
  - Institut Sainte-Catherine, Avignon
  - CHU Bordeaux - Hôpital Saint-André, Bordeaux
  - Polyclinique de Bordeaux Nord, Bordeaux
  - CHRU Brest - Hôpital Morvan, Brest
  - Centre François Baclesse, Caen
  - CHIC Créteil, Créteil
  - Centre Guillaume le Conquérant, Le Havre
  - Centre Hospitalier Bretagne Sud, Lorient
  - Centre Léon Bérard, Lyon
  - AP-HM La Timone Adultes, Marseille
  - Centre Antoine Lacassagne, Nice
  - CHU Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Pôle Hospitalier Mutualiste- Centre Etienne Dolet, Saint-Nazaire
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Strasbourg Oncologie Libérale, Strasbourg
  - Hopitaux du Léman, Thonon-les-Bains
  - Clinique Pasteur Bâtiment l'Atrium, Toulouse
  - Institut Claudius Regaud, Toulouse
  - CHU TOURS (Hôpital Bretonneau), Tours
  - Centre de Radiothérapie Marie Curie, Valence
  - Institut de Cancérologie de lorraine (ICL), Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Bernier J, Domenge C, Ozsahin M, Matuszewska K, Lefebvre JL, Greiner RH, Giralt J, Maingon P, Rolland F, Bolla M, Cognetti F, Bourhis J, Kirkpatrick A, van Glabbeke M; European Organization for Research and Treatment of Cancer Trial 22931. Postoperative irradiation with or without concomitant chemotherapy for locally advanced head and neck cancer. N Engl J Med. 2004 May 6;350(19):1945-52. doi: 10.1056/NEJMoa032641. PMID 15128894
- [Background] Seiwert, TC, clement, P. M, Del Campo, J, de Mont-Serrat, H., Thurm, H. C., Blackman, A. S., and Cohen, E. E. BIBW 2992 versus cetuximab in patients with metastatic or recurrent head and neck cancer (SCCHN) after failure of platinum-containing therapy with a cross-over period for progressing patients: Preliminary results of a randomized, open-label phase II study. Journal of Clinical Oncology 28(15 suppl). 2010.
- [Background] Cooper JS, Pajak TF, Forastiere AA, Jacobs J, Campbell BH, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Machtay M, Ensley JF, Chao KS, Schultz CJ, Lee N, Fu KK; Radiation Therapy Oncology Group 9501/Intergroup. Postoperative concurrent radiotherapy and chemotherapy for high-risk squamous-cell carcinoma of the head and neck. N Engl J Med. 2004 May 6;350(19):1937-44. doi: 10.1056/NEJMoa032646. PMID 15128893
- [Background] Carpenter G, Cohen S. Epidermal growth factor. J Biol Chem. 1990 May 15;265(14):7709-12. No abstract available. PMID 2186024
- [Background] Mendelsohn J. Epidermal growth factor receptor inhibition by a monoclonal antibody as anticancer therapy. Clin Cancer Res. 1997 Dec;3(12 Pt 2):2703-7. PMID 10068277
- [Background] Salomon DS, Brandt R, Ciardiello F, Normanno N. Epidermal growth factor-related peptides and their receptors in human malignancies. Crit Rev Oncol Hematol. 1995 Jul;19(3):183-232. doi: 10.1016/1040-8428(94)00144-i. No abstract available. PMID 7612182
- [Background] Grandis JR, Tweardy DJ. TGF-alpha and EGFR in head and neck cancer. J Cell Biochem Suppl. 1993;17F:188-91. doi: 10.1002/jcb.240531027. PMID 8412192
- [Background] Baselga J. New therapeutic agents targeting the epidermal growth factor receptor. J Clin Oncol. 2000 Nov 1;18(21 Suppl):54S-9S. No abstract available. PMID 11060328
- [Background] Fan Z, Mendelsohn J. Therapeutic application of anti-growth factor receptor antibodies. Curr Opin Oncol. 1998 Jan;10(1):67-73. doi: 10.1097/00001622-199801000-00011. PMID 9466487
- [Background] Milas L, Mason K, Hunter N, Petersen S, Yamakawa M, Ang K, Mendelsohn J, Fan Z. In vivo enhancement of tumor radioresponse by C225 antiepidermal growth factor receptor antibody. Clin Cancer Res. 2000 Feb;6(2):701-8. PMID 10690556
- [Background] Kaplan EL and Meier P. Nonparametric estimation from incomplete observations. J Am Stat Assoc 1958; 53: 457-81. 2006.
- [Background] Gregoire V, Eisbruch A, Hamoir M, Levendag P. Proposal for the delineation of the nodal CTV in the node-positive and the post-operative neck. Radiother Oncol. 2006 Apr;79(1):15-20. doi: 10.1016/j.radonc.2006.03.009. Epub 2006 Apr 17. PMID 16616387
- [Background] Lapeyre M, Henrot P, Alfonsi M, Bardet E, Bensadoun RJ, Dolivet G, Favrel V, Gallocher O, Giraud P, Graff P, Guerif S, Lagarde P, Lartigau E, Marchesi V, Pommier P, Rives M, Tortochaux J, Toussaint B, Verrelle P, Bourhis J, Calais G; Groupe Oncologie Radiotherapie Tete et Cou. [Propositions for the selection and the delineation of peritumoral microscopic disease volumes in oral cavity and oropharyngeal cancers (lymph nodes excluded)]. Cancer Radiother. 2005 Jun;9(4):261-70. doi: 10.1016/j.canrad.2005.03.005. Epub 2005 Apr 25. French. PMID 16081023
- [Background] Gregoire V, Levendag P, Ang KK, Bernier J, Braaksma M, Budach V, Chao C, Coche E, Cooper JS, Cosnard G, Eisbruch A, El-Sayed S, Emami B, Grau C, Hamoir M, Lee N, Maingon P, Muller K, Reychler H. CT-based delineation of lymph node levels and related CTVs in the node-negative neck: DAHANCA, EORTC, GORTEC, NCIC,RTOG consensus guidelines. Radiother Oncol. 2003 Dec;69(3):227-36. doi: 10.1016/j.radonc.2003.09.011. PMID 14644481
- [Background] Prescribing, Recording, and Reporting Intensity-Modulated Photon-Beam Therapy (IMRT)(ICRU Report 83) ICRU Report 83, Journal of the ICRU Vol. 10 No. 1. 2011.
- [Background] Chao KS, Majhail N, Huang CJ, Simpson JR, Perez CA, Haughey B, Spector G. Intensity-modulated radiation therapy reduces late salivary toxicity without compromising tumor control in patients with oropharyngeal carcinoma: a comparison with conventional techniques. Radiother Oncol. 2001 Dec;61(3):275-80. doi: 10.1016/s0167-8140(01)00449-2. PMID 11730997
- [Derived] Racadot S, Thennevet I, Ouldbey Y, Kaminsky MC, Bosset M, Martin L, Tao Y, Sire C, de Raucourt D, Alfonsi M, Malaurie E, Tourani JM, Fournel P, Vauleon E, Modesto A, Rolland F, Metzger S, Pommier P, Chabaud S, Dussart S; GORTEC group. Afatinib maintenance therapy following post-operative radiochemotherapy in head and neck squamous cell carcinoma: Results from the phase III randomised double-blind placebo-controlled study BIB2992ORL (GORTEC 2010-02). Eur J Cancer. 2023 Jan;178:114-127. doi: 10.1016/j.ejca.2022.10.023. Epub 2022 Nov 9. PMID 36434888